CLINICAL TRIAL: NCT03330860
Title: Effectiveness of 12 Clips in Maternal and Neoanatal Health Through Applied Neuroscience Tools (Neuromarketing Strategy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Capsule1
Record Dates: First submitted 2015-11-19; First posted 2017-11-06 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy

STUDY DESIGN:
Intervention Model Description: Crossover randomized clinical trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromarketing strategy (Experimental): Twelve clips regarding maternal and neonatal health topics, designed with mixed 2D and 3D elements, each one about 45 seconds long (prepared based on the best available evidence and validated by clinical experts).
  Interventions: Other: Twelve clips regarding maternal and neonatal health topics
- No-capsule group (Active Comparator): Control clip with 2D elements about 45 seconds long, containing information on prenatal control and presented in conventional format (narration, static images and on screen text).
  Interventions: Other: Control Clip

INTERVENTIONS:
Other: Twelve clips regarding maternal and neonatal health topics — Twelve clips regarding maternal and neonatal health topics, designed with mixed 2D and 3D elements, each one about 45 seconds long (prepared based on the best available evidence and validated by clinical experts).
  Arms: Neuromarketing strategy
Other: Control Clip — Control clip with 2D elements about 45 seconds long, containing information on prenatal control and presented in conventional format (narration, static images and on screen text).
  Arms: No-capsule group

SUMMARY:
Objective: To evaluate the effectiveness of 12 knowledge transfer clips of maternal and neonatal health in order to generate knowledge appropriation. Methodology: Randomized cross-over clinical trial with a non-probabilistic sample of intentional feature of 150 subjects: pregnant women, non-pregnant women and men. Participants will be evaluated during the observation of 13 clips (one of them is the control clip) in which sequence will be assigned randomly. The level of attention will be assessed by means of eye tracking, to see the ocular gaze and fixation in relation to the content of clips, and emotional reaction through the psychophysiological record (galvanic skin response). In addition, recall of information will be assessed through the application of questionnaires at the end of each video. The analysis will focus on identifying differences in the three outcomes between intervention clips and the control clip, and between the three groups, and determine the clips and segments that generate greater emotional response, attention and recall.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, Men, and Non-pregnant women that accept to participate in the study

Exclusion Criteria:

* Participant that don't sign informed consent or have clinically significant visual or auditory impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Emotional impact (electrodermal activity) | 1 day
  Monitoring of autonomous activity will be carried out through the registration of electrodermal activity (galvanic skin response), which allows the evaluation of emotional reaction. Electrodermal activity will be measured by a computerized psychophysiological recording equipment. The electrodes will be placed in the distal phalanx of the third and fourth finger of the non-dominant hand with SE-35 sensors connected to a T-601 preamplifier (J & J Enterprises Seattle, WA).
  The analysis of skin conductance will be carried out with the amplitude of electrodermal response which is obtained by the subtraction of the lowest conductance of the latency period from the peak conductance. This analysis will be performed for each event identified in each clip for each subject.

SECONDARY OUTCOMES:
Recall (Questionnarie) | 1 day
  The measurement of the recall component will be carried out by filling out a knowledge test in form of questionnaire once the screening of each video has finished. The proportion of correct answers by questionnaire will be calculated.
Attention (Eye tracking) | 1 day
  The eye tracking method will be applied to evaluate the attention to the visual stimulus of the clips. By means of the Eye Tracker Tobii Tx300 tracking equipment, the eye movements will be recorded. The record of how and when gaze is focused on the areas of interest (AOIs) will be measured with the following variables: 1. Duration until the first fixation in an AOI (Time to First Fixation - TFF) in seconds, and number of fixations before focusing on an AOI (Fixations Before - FB). These two measures indicate the anticipation with which attention is fixed in a specific area of the screen. 2. Duration and number of all fixations made in an AOI. These measurements indicate the duration of the fixation in each AOI and the number of times the participant fixes his gaze on that area.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional de Colombia, Bogotá, Colombia